CLINICAL TRIAL: NCT06969196
Title: Artificial Intelligence-Generated Written Communication for Families of Intensive Care Unit Patients - A Pilot Study
Brief Title: Artificial Intelligence-Generated Written Communication for Families of Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25040406
Record Dates: First submitted 2025-04-18; First posted 2025-05-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Communication; ICU
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Written Communication (Experimental): AI-edited, ICU clinician edited written communication
  Interventions: Other: Written Communicatoin

INTERVENTIONS:
Other: Written Communicatoin — ICU clinicians will be asked to edit AI-generated written summaries for content and clarity before they are delivered to families

SUMMARY:
Our research group has developed an approach for providing families of ICU patients with daily written summaries of care as a supplement to traditional verbal communication. Written summaries describe the patient's main ICU problems and management plan and are delivered to families each day. Despite the benefits of written communication to both the family and clinician experience, the main barrier to implementing this communication approach is the time required for clinicians to create a written summary. For the proposed pilot study, the investgators will ask ICU clinicians to identify patients and respective families for whom there has been a challenge with communication. The investigators will ask ICU clinicians to edit AI-generated written summaries for content and clarity before they are delivered to families. The investigators hypothesize that this process will acceptable and feasible for ICU clinicians and families.

ELIGIBILITY:
Surrogate Inclusion

* One self-identified adult decision maker for an adult medical ICU patient cared for on the 10W ICU
* Member of the primary ICU team believes the respective patient will require at least three additional days of ICU care
* Member of the primary ICU team has identified at least one communication challenge with the patient's surrogate(s) including but not limited to:

  1. Complex medical issues requiring frequent updates to families
  2. Complex family dynamics (i.e., multiple involved family members)
  3. Increased anxiety/stress of surrogate(s)
  4. Difficult to provide updates to family members because they do not visit ICU regularly or are hard to reach by phone

Surrogate Exclusion

* Surrogate cannot read or understand English
* Surrogate is unwilling or unable to participate in study procedures
* Patient is decisional and refuses to allow surrogate participation

Clinician Inclusion • Advanced practice provider (APP) on the medical ICU team on the 10W ICU

Clinician Exclusion

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Communication Quality (Clinicians) | Through study completion, an average of one week
  Clinician participants will ratings of quality of AI-generated written summaries and whether written summaries address family-specific communication challenges (5-point Likert scale, 1-5 points with higher scores indicating better quality)
Communication Quality (Families/Surrogates) | Average one week after enrollment
  The Family Inpatient Communication Survey (FICS) is a 30-item survey measuring of the quality of communication with the treatment team from the perspective of families of hospitalized patients. Items on this survey measure the informational and emotional aspects of communication, and each item of this survey is rated on a 5-point Likert scale from strongly agree to strongly disagree (30-150 points with higher scores indicating better quality communication)
Acceptability of intervention | Average one week after enrollment
  Acceptability of the intervention will reflected in adequate enrollment and an average score of at least 3.5 on surveys with 5-point Likert scale measures including the Acceptability of Intervention (AIM), Appropriateness of Intervention (IAM), and Feasibility of Intervention Survey (FIM) (1-5 point with higher scores being better)
Feasibility of intervention | Through study completion, an average of one week
  Feasibility will be determined by written communication being created for at least 80% of all ICU days and less than 5 minutes on average being spent editing each AI-generated summary.

OTHER OUTCOMES:
Analysis of Individual Interviews | Average one week after enrollment
  Individual interviews will be conducted by a study investigator using an interview guide Interviews will last approximately 15 minutes. Interviews will be transcribed and coded. Themes identified in qualitative analysis will be used to inform and provide explanations for quantitative results.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JJ, Mathur S, Gerhart J, Glover CM, Ritz E, Basapur S, Greenberg JA. Written communication and the ICU team experience (WRITE): A pre-post intervention study. Intensive Crit Care Nurs. 2024 Oct;84:103753. doi: 10.1016/j.iccn.2024.103753. Epub 2024 Jun 25. PMID 38924848
- [Background] Greenberg JA, Basapur S, Quinn TV, Bulger JL, Schwartz NH, Oh SK, Ritz EM, Glover CM, Shah RC. Daily Written Care Summaries for Families of Critically Ill Patients: A Randomized Controlled Trial. Crit Care Med. 2022 Sep 1;50(9):1296-1305. doi: 10.1097/CCM.0000000000005583. Epub 2022 May 23. PMID 35607975
- [Background] Bulger JL, Quinn TV, Glover CM, Basapur S, Shah RC, Greenberg JA. Written Care Summaries Facilitate Communication Between Families and Providers of ICU Patients: A Pilot Study. Crit Care Explor. 2021 Jul 13;3(7):e0473. doi: 10.1097/CCE.0000000000000473. eCollection 2021 Jul. PMID 34278309